CLINICAL TRIAL: NCT00206089
Title: The "EXTEND" Study: A Randomized, Double-blind, Parallel-group, Phase III b, Multi-centre Study Evaluating Extended Prophylactic Treatment With Melagatran/Ximelagatran Versus Enoxaparin for the Prevention of Venous Thromboembolic Events in Patients Undergoing Elective Hip Replacement or Hip Fracture Surgery.
Brief Title: Melagatran/Ximelagatran Versus Enoxaparin for the Prevention of Venous Thromboembolic Events
Acronym: EXTEND
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Melagatran/ximelagatran was withdrawn from the market and clinical development in February 2006 in the interest of patient safety.
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D4003C00030
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Thromboembolism
Keywords: Prevention of venous thromboembolic events in patients undergoing elective hip replacement or hip fracture surgery
MeSH Terms: conditions — Thromboembolism | interventions — ximelagatran; melagatran

INTERVENTIONS:
Drug: EXANTA
  Other Names: Melagatran/Ximelagatran

SUMMARY:
This study is being carried out to study the efficacy and safety of treatment with melagatran injection followed by ximelagatran tablets in preventing blood clots, compared with enoxaparin for a period of 5-6 weeks. A separate visit, independent from the study will be done approximately 6 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Female or male aged 18 years and over
* Patient scheduled for primary elective hip replacement or patient requiring surgery for hip fracture.

Exclusion Criteria:

* History of heparin-induced thrombocytopenia
* Conditions associated with increased risk of bleeding, renal impairment, known active liver disease or liver insufficiency.
* Myocardial infarction, Ischemic stroke or Transient Ischemic Attack (TIA), systemic embolism or venous thrombo-embolism within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300
Dates: Start 2005-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Non-inferiority for the prevention of VTE or VTE related death

SECONDARY OUTCOMES:
Superiority regarding major bleeding or the percentage of patients requiring donor blood transfusion.
Safety

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Medical Science Director, MD, Study Director — AstraZeneca
Locations (125):
- Austria (9):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Leoben
  - Research Site, Neunkirchen
  - Research Site, Neustadt
  - Research Site, Sankt Johann in Tirol
  - Research Site, Viborg
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Denmark (10):
  - Research Site, Aarhus
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Herlev
  - Research Site, Hillerød
  - Research Site, Holstebro
  - Research Site, Hvidovre
  - Research Site, Hørsholm
  - Research Site, Silkeborg
  - Research Site, Vejle
- Finland (6):
  - Research Site, Hus
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Oys
  - Research Site, Tampere
  - Research Site, Turku
- France (9):
  - Research Site, Amiens
  - Research Site, Annecy
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Saint-Etienne
- Germany (9):
  - Research Site, Bad Mergentheim
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Garmisch-Partenkirchen
  - Research Site, Halle
  - Research Site, Rheinfelden
  - Research Site, Sommerfeld
  - Research Site, Wiesbaden
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Gyzr
  - Research Site, Kecskemét
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Székesthérvár
- Mexico (3):
  - Research Site, Estado de México
  - Research Site, Guadalajara
  - Research Site, Mexico City
- Netherlands (8):
  - Research Site, Assen
  - Research Site, Breda
  - Research Site, Groningen
  - Research Site, Hilversum
  - Research Site, Leeuwarden
  - Research Site, Sittard
  - Research Site, Zaandam
  - Research Site, Zwolle
- Norway (17):
  - Research Site, Ålesund
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Drammen
  - Research Site, Elverum
  - Research Site, Gjettum
  - Research Site, Hagavik
  - Research Site, Kongsberg
  - Research Site, Kongsvinger
  - Research Site, Larvik
  - Research Site, Levanger
  - Research Site, Lillehammer
  - Research Site, Nordbyhagen
  - Research Site, Oslo
  - Research Site, Skien
  - Research Site, Stavanger
  - Research Site, Trondheim
- Poland (8):
  - Research Site, Biaystok
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Gdansk
  - Research Site, Lublin
  - Research Site, Od
  - Research Site, Warsaw
  - Research Site, Wrocraw
- Portugal (7):
  - Research Site, Barreiro
  - Research Site, Cascais
  - Research Site, Lisbon
  - Research Site, Parede
  - Research Site, Setúbal
  - Research Site, Torres Vedras
  - Research Site, Vila Franca de Xira
- South Africa (3):
  - Research Site, Durban
  - Research Site, Gauteng
  - Research Site, Sandton
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Ourense
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (15):
  - Research Site, Borås
  - Research Site, Falköping
  - Research Site, Falun
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Kalmar
  - Research Site, Kungälv
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Mölndal
  - Research Site, Örebro
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Uddevalla
  - Research Site, Uppsala
- Switzerland (6):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lugano
  - Research Site, Luzem
  - Research Site, Zurich

REFERENCES:
- [Derived] Agnelli G, Eriksson BI, Cohen AT, Bergqvist D, Dahl OE, Lassen MR, Mouret P, Rosencher N, Andersson M, Bylock A, Jensen E, Boberg B; EXTEND Study Group. Safety assessment of new antithrombotic agents: lessons from the EXTEND study on ximelagatran. Thromb Res. 2009;123(3):488-97. doi: 10.1016/j.thromres.2008.02.017. Epub 2008 May 15. PMID 18485453